CLINICAL TRIAL: NCT03402074
Title: Group Hypnosis for Stress Reduction - a Feasibility Study
Brief Title: Group Hypnosis for Stress Reduction
Acronym: Hypnostress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Benno Brinkhaus, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hypnostress
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Hypnosis (Experimental): 5 sessions of group hypnosis, each 90 minutes; plus CDs/MP3 recordings to train at home
  Interventions: Behavioral: Group hypnosis

INTERVENTIONS:
Behavioral: Group hypnosis — 5 session of group hypnosis, each 90 minutes, to reduce subjective stress and increase relaxation. Additional auditapes of hypnosis sessions as hoemwork

SUMMARY:
This prospective feasibility study aims to test a 5 week group hypnosis training as intervention to reduce perceived psychological stress in healthy subjects.

DETAILED DESCRIPTION:
In a pre- post comparison the feasibility of a standardized weekly 90 minutes group hypnosis training including CDs/MP3 recordings as homework to reduce perceived psychological stress in healthy subjects is investigated. Outcomes are measured quantitatively and qualitatively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or health-stable participants between 18 and 70 years with subjective increased intensity of stress in the last four weeks on the visual analogue scale rated between 40 -100 mm (VAS 0 - 100 mm)
* Ability to consent and sign declaration of informed consent

Exclusion Criteria:

* Current or planned participation in a stress management program within the next 17 weeks
* Current use of psychotherapeutic treatment
* presence of moderate or severe acute or chronic disease
* presence of an acute or chronic mental disorder
* Participation in a study within the last 2 months prior to enrollment
* Lack of understanding of the German language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress on Visual Analogue Scale | 5 weeks
  VAS 0-100 mm
Cohens Perceived Stress Scale 10 Items | 5 weeks
Likert-Skala | 5 weeks
  about stressreduction
ADS-K (Depression) | 5 weeks
General Self Efficacy Scale (Schwarzer) | 5 weeks
SF 36 Quality of Life | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hochschulambulanz für Naturheilkunde, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided